CLINICAL TRIAL: NCT06258564
Title: The Adjuvant Effect of HPV Vaccination on Recurrence of Cervical Intraepithelial Neoplasia Grade 2 or Worse in Women Undergoing Conization: Retrospective Cohort Study
Brief Title: The Adjuvant Effect of HPV Vaccination on Recurrence of Cervical Precancer or Carcinoma in Women Undergoing Conization
Status: Completed | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Sponsor
Other Study IDs: PAVIVE2024; Cooperatio 31 fund (Other Grant/Funding Number: Charles University, Prague)
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-01

CONDITIONS: Cervical Intraepithelial Neoplasia Grade 2/3; Recurrence
Keywords: HPV; vaccination; CIN2+ recurrence; conization
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- single cohort of women with cervical excision for CIN2+: single cohort of women with cervical excision for CIN2+; those with HPV vaccination and those without HPV vaccination
  Interventions: Biological: vaccination against human papillomavirus infection (HPV vaccination)

INTERVENTIONS:
Biological: vaccination against human papillomavirus infection (HPV vaccination) — Women with or without HPV vaccination before or after excision

SUMMARY:
Assessment of the association between human papillomavirus vaccination (HPV) and recurrences of cervical intraepithelial neoplasia grade 2 or worse (CIN2+) in women undergoing conization.

DETAILED DESCRIPTION:
The implementation of vaccination against human papillomavirus (HPV) in the national immunization program for the young age cohort was subsequently extended to previously unvaccinated adult women who underwent conization due to cervical intraepithelial neoplasia grade 2 or worse (CIN2+).

These women are offered HPV vaccination, often completed post-excision. Observational and clinical studies conducted between 2010 and 2023 have demonstrated that HPV vaccination contributes to a >70% reduction in CIN2+ recurrence in women after conization. However, the outcomes of these studies have not conclusively shown whether the adjuvant effect of HPV vaccination depends on the vaccine type (bi-, quadri-, or nona-valent), the timing and completeness of vaccination, and other factors.

This study aims to assess the mentioned factors and potentially reveal new ones, such as age, health status, etc. It is planned to be conducted using the laboratory records of women who underwent conization between 2010 and 2024, with their cervical screening examinations performed at the central laboratory UNILABS in Prague

ELIGIBILITY:
Inclusion Criteria:

* Women >18 years, with conization for CIN2+ (HSIL)
* Women who had more than one examination during a follow-up period of >6 months.

Exclusion Criteria:

- Women who underwent hysterectomy after conization.

* Women who had excision procedures other than cervical excision.
* Women who did not undergo any other cytological/histological examinations.
* Women with more than one conization before CIN2+ recurrence

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population consists of women who underwent conization for CIN2+, and the laboratory examination of conization and other samples was conducted at the central laboratory of UNILABS. The follow-up period for the population must be at least 6 months, with at least one negative finding before a recurrence of CIN2+ is identified.
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
CIN2+ recurrence rate | 2010-2024
  CIN2+ recurrence rate - obtained from the number of women with this find-ing related the number of women with no finding within the time period since the conization; The recurrence rate of CIN2+ will be assessed in relation to vaccination, vaccine type, vaccination completeness, etc., using specific uni-variate analysis (incidence rate ratio) and multivariate analysis (incidence rate ratio or hazard ratio, as appropriate)

SECONDARY OUTCOMES:
CIN2+ recurrence frequency | 2010-2024
  CIN2+ recurrence frequency - percentage proportion of women with this finding related to all women in follow-up; The recurrence frequency of CIN2+ will be assessed in relation to vaccination, vaccine type, vaccination completeness, etc., using specific univariate analysis (odds ratio, relative risk) and multivariate analysis (odds ratio, relative risk, as appropriate)

CONTACTS AND LOCATIONS:
Overall Officials: Marek Petráš, assoc.prof., Principal Investigator — Department of Epidemiology and Biostatistics, Third Faculty of Medicine, Charles University, Prague, Czech Republic
Locations (2):
- Czechia (2):
  - Department of Epidemiology and Biostatistics, Third Faculty of Medicine, Charles University, Prague
  - Unilabs Pathology K.S, Prague

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petras M, Dvorak V, Lomozova D, Macalik R, Neradova S, Dlouhy P, Malinova J, Rosina J, Lesna IK. Timing of HPV vaccination as adjuvant treatment of CIN2+ recurrence in women undergoing surgical excision: a meta-analysis and meta-regression. Sex Transm Infect. 2023 Dec;99(8):561-570. doi: 10.1136/sextrans-2023-055793. Epub 2023 Aug 8. PMID 37553234
- See also: Timing of HPV vaccination as adjuvant treatment of CIN2+ recurrence in women undergoing surgical excision: a meta-analysis and meta-regression — https://sti.bmj.com/content/99/8/561